CLINICAL TRIAL: NCT03619863
Title: A Natural History Cohort Study of the Safety, Effectiveness, and Practice of Treatment for People With Hemophilia
Brief Title: ATHN 7: Hemophilia Natural History Study
Acronym: ATHN 7
Status: Completed | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN 7
Record Dates: First submitted 2018-07-25; First posted 2018-08-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A With Inhibitor; Haemophilia A Without Inhibitor; Hemophilia B With Inhibitor; Haemophilia B Without Inhibitor
Keywords: Hemophilia; Non-Factor Products; Bypassing Agents; Clotting Factor Replacement Products
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a real-world study of the safety of the treatments used for people with hemophilia. The study will follow people with hemophilia A or B from across the country for about 4 years as they receive treatment. The hemophilia treatment center (HTC) physician and participant will decide on the FDA-approved treatment to be used which may include non-factor products, bypassing agents, or clotting factor replacement products. The goal of this research is to study the use of hemophilia treatment products and their outcomes.

DETAILED DESCRIPTION:
This non-interventional, minimal risk cohort study will enroll and follow patients with hemophilia A or B as they receive hemophilia treatment for 4 years. This is a pragmatic study of real-world practices across a wide range of patients which will be ongoing as new treatment products receive FDA approval and will be advantageous to the entire hemophilia community. The total study duration is planned for 6 years.

The patients are seen at baseline, annually, and at study exit. Patients will also receive routine quarterly follow-up phone calls from HTC staff to review medical history, bleed events, and product treatment history. Other visits for unplanned events or for the change of treatment product will be scheduled as necessary. All required study visits will be planned to coincide with routine clinical care whenever possible. Co-enrollment in the ATHNdataset by patients is required to participate in the study.

Please note - the treatment regimen will be at the discretion of the patients' hemophilia caregivers. No treatment products are being provided by the study nor will the participants be paid. However, inhibitor titer testing will be provided at no cost to patients by the Center for Disease Control and Prevention (CDC).

The primary objective is to determine the safety of non-factor products, bypassing agents or clotting factor replacement products when used for people with hemophilia with or without inhibitors. Safety will be measured by those events listed in the European Haemophilia Safety Surveillance (EUHASS).

Data collected will include eligibility, demographics, medical history, hemophilia history (genotype and family history), inhibitor history and immune tolerance induction (ITI) treatment regimen (if applicable), co-morbidities at baseline (i.e., HIV, Hepatitis C), detailed treatment product(s) usage, bleeding events, surgical procedures, and EUHASS adverse events and other adverse events of special interest. Data collection will also include patient-reported outcome questionnaires regarding health-related quality of life, treatment use and patient perceptions of treatment products.

Sub-studies

A number of sub-studies are planned with pharmaceutical sponsors to collect information from patients about their specific product use. Participation in these sub-studies (Product Specific Modules) is optional and sub-study visits will be planned to coincide with HTC visits. The modules will collect information from patients about their perception and use of treatment products, physical activity levels and other general health questions. This data will be collected via questionnaire.

Data Collection System

All data collected will be entered into electronic case report forms (eCRFs) within the secure ATHN System by HTC site personnel. All participating study sites will have in place a current, executed Data Use and Business Associate Agreement (DUBAA) with ATHN.

ELIGIBILITY:
Inclusion Criteria:

1. Congenital hemophilia A or B of any severity with or without inhibitors receiving a current therapy, a non-factor product, or for whom use of a non-factor product is a possibility;
2. Able to give informed consent (by patient or parent/authorized guardian); and
3. Co-enrollment in the ATHNdataset.

Exclusion Criteria:

1. Presence of any known bleeding disorder other than congenital hemophilia A or B;
2. Presence of concurrent hemophilia and a second hemostatic defect (low Von Willebrand Factor (VWF) without Von Willebrand disease (VWD) diagnosis is not excluded); and
3. Unable or unwilling to comply with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll approximately 280 patients with hemophilia who meet the eligibility criteria and receiving care from one of the ATHN-affiliated Hemophilia Treatment Centers (HTC).
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Safety of treatment products used for hemophilia care will be assessed based on the number of reportable European Haemophilia Safety Surveillance (EUHASS) events documented on the ATHN Adverse Event Module Form. | 6 years
  All treatment-related reportable adverse events will be documented on the ATHN Adverse Event Module Form based on EUHASS reportable events which include: death, factor inhibitor development, venous thrombosis, allergic reactions, treatment-emergent side effects, new malignancies, cardiovascular events, and blood-borne infections. Other treatment-related events to be documented on the ATHN Adverse Event Module Form including thrombotic microangiopathies, injection site reactions, drug-induced liver injury and anti-drug antibodies.

SECONDARY OUTCOMES:
Effectiveness of non-factor products, bypassing agents and clotting factor replacement products will be evaluated based on the participant's number of bleeding events reported as the annualized bleeding rate (ABR). | 6 years
  Annualized bleeding rates (bleeds/year) are calculated as the number of bleeding events divided by length of time of the treatment regimen, in years. Participants will report bleeding including spontaneous bleeding, traumatic bleeding, joint related and non-joint bleeding during routine quarterly follow-up with hemophilia care providers. Participants will also have blood loss associated with surgical procedures documented through medical chart review as noted by the surgical care providers. All bleeding data will be gathered and reported.
Dosing regimens for hemophilia treatment products and total amount utilized by the study participant for prophylaxis and treatment of bleeds will be assessed. | 6 years
  The routine quarterly contact by hemophilia care providers with study participants will be used to evaluate their treatment use and will document dosing regimens of hemophilia treatment products, amount of product used, number of participants switching to a different product, number of participants switching between factor and non-factor products, and/or number of participants staying on the current treatment product and the reason for their choice of treatment.
Target joint monitoring | 6 years
  The number and location of target joints at study entry, incidence of target joint development while on study, and the number of target joints that resolve following study enrollment will be documented and analyzed.
  The number and location of target joints at study entry, incidence of target joint development while on study, and the number of target joints that resolve following study enrollment will be documented and analyzed.
Efficacy of treatment is rated by health-related outcomes tools: EQ-5D-5L, Patient-Reported Outcomes Measurement Information System (PROMIS), Global Adherence Rating (GAR), and Treatment Satisfaction with Medicines Questionnaire (SATMED-Q). | 6 years
  EuroQol Group's EQ-5D-5L assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Opinions in the 5 categories can be stated as a health profile or converted to a single summary index number. Opinion on overall health is on a scale of 0 to 100 with 100 as best health imagined. PROMIS Profile 29 (adults)/ 25 (peds)/ Parent Proxy 25 assess physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles/activities, and pain. Questions are ranked on a 5-point Likert Scale and one question on pain has a 11-point rating scale. GAR assesses adherence to the prescribed regimen on a scale of 0 to 10 with 10 always taken as prescribed. SATMED-Q assesses the satisfaction with the prescribed treatment based on a Likert scale and provides a total score for treatment satisfaction by summing all domains: side effects, efficacy, convenience and ease of use, impact of the medicine, medical follow-up/review and overall opinion.
Real world effectiveness of treatment products assessed by the healthcare providers as measure by the number and types of medical visits and/or hospitalizations per year. | 6 years
  Healthcare providers will document the number and types of medical visits/hospitalization per year that are related to hemophilia care and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Buckner, MD, MSc, Principal Investigator — Hemophilia and Thrombosis Center/ University of Colorado Anschutz Medical Campus; Michael Recht, MD, PhD, Principal Investigator — The Hemophilia Center at Oregon Health & Science University
Locations (29):
- United States (29):
  - Arizona Hemophilia and Thrombosis Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Orthopaedic Institute for Children HTC, Los Angeles, California
  - Orthopedic Institute for Children Hemophilia Program, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Hemophilia and Thrombosis Center/ University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida Hemophilia Treatment Center, Gainesville, Florida
  - Comprehensive Bleeding Disorders Center at Emory University and Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center (IHTC), Indianapolis, Indiana
  - Louisiana Center for Bleeding and Clotting Disorders, Tulane University, New Orleans, Louisiana
  - Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - Massachusetts General Hospital Comprehensive Hemophilia and Thrombosis Treatment Center, Boston, Massachusetts
  - Michigan State University Center for Bleeding and Clotting Disorders, East Lansing, Michigan
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - The John Bouhasin Center for Children with Bleeding Disorders, St Louis, Missouri
  - Hemostasis and Thrombosis Center of Nevada, Las Vegas, Nevada
  - Hemostasis and Thrombosis Center of Nevada, Reno, Nevada
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Wake Forest University Health Science, Winston-Salem, North Carolina
  - Northwest Ohio Hemophilia Treatment Center at the Toledo Hospital, Toledo, Ohio
  - The Hemophilia Center at Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Penn Comprehensive Hemophilia and Thrombophilia Program/Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - The Center for Cancer and Blood Disorders, Children's Medical Center of Dallas, Dallas, Texas
  - Gulf States Hemophilia and Thrombosis Center, Houston, Texas
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin

REFERENCES:
- [Background] Ragni MV. Targeting Antithrombin to Treat Hemophilia. N Engl J Med. 2015 Jul 23;373(4):389-91. doi: 10.1056/NEJMcibr1505657. No abstract available. PMID 26200986
- [Background] Gouw SC, van den Berg HM, Fischer K, Auerswald G, Carcao M, Chalmers E, Chambost H, Kurnik K, Liesner R, Petrini P, Platokouki H, Altisent C, Oldenburg J, Nolan B, Garrido RP, Mancuso ME, Rafowicz A, Williams M, Clausen N, Middelburg RA, Ljung R, van der Bom JG; PedNet and Research of Determinants of INhibitor development (RODIN) Study Group. Intensity of factor VIII treatment and inhibitor development in children with severe hemophilia A: the RODIN study. Blood. 2013 May 16;121(20):4046-55. doi: 10.1182/blood-2012-09-457036. Epub 2013 Apr 3. PMID 23553768
- [Background] Shima M, Hanabusa H, Taki M, Matsushita T, Sato T, Fukutake K, Fukazawa N, Yoneyama K, Yoshida H, Nogami K. Factor VIII-Mimetic Function of Humanized Bispecific Antibody in Hemophilia A. N Engl J Med. 2016 May 26;374(21):2044-53. doi: 10.1056/NEJMoa1511769. PMID 27223146
- [Background] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557
- [Background] Carr ME, Tortella BJ. Emerging and future therapies for hemophilia. J Blood Med. 2015 Sep 3;6:245-55. doi: 10.2147/JBM.S42669. eCollection 2015. PMID 26366108
- [Background] Sehgal A, Barros S, Ivanciu L, Cooley B, Qin J, Racie T, Hettinger J, Carioto M, Jiang Y, Brodsky J, Prabhala H, Zhang X, Attarwala H, Hutabarat R, Foster D, Milstein S, Charisse K, Kuchimanchi S, Maier MA, Nechev L, Kandasamy P, Kel'in AV, Nair JK, Rajeev KG, Manoharan M, Meyers R, Sorensen B, Simon AR, Dargaud Y, Negrier C, Camire RM, Akinc A. An RNAi therapeutic targeting antithrombin to rebalance the coagulation system and promote hemostasis in hemophilia. Nat Med. 2015 May;21(5):492-7. doi: 10.1038/nm.3847. Epub 2015 Apr 13. PMID 25849132
- [Derived] Buckner TW, Carpenter SL, Daoud N, Kempton CL, Lee L, Malec L, McLean TW, Morton P, O'Neill C, Staber JM, Wang M, Croteau SE, Recht M. Safety and Effectiveness of Emicizumab in People With Haemophilia A Enrolled in the ATHN 7 Haemophilia Natural History Study. Haemophilia. 2025 Nov 11. doi: 10.1111/hae.70151. Online ahead of print. PMID 41220279